CLINICAL TRIAL: NCT06159517
Title: Post-Market Clinical Follow-up Registry to Evaluate the Safety and Performance of the HL 40 Heart Lung Machine and the Temperature Probes in Patients Undergoing Cardiac / Thoracic / Vascular Surgery
Brief Title: Heart Lung Machine Registry
Acronym: HeaLMe
Status: Terminated | Type: Observational
Why Stopped: The index device HL 40 has been discontinued
Sponsor: Maquet Cardiopulmonary GmbH (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Other Study IDs: 3110158
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Surgery; Thoracic Surgery; Vascular Surgery; Cardiopulmonary Bypass
Keywords: Heart Lung Machine; HL 40; Temperature Probes; TPO-D-HLM L1.8 Adult; TPO-D-HLM L1.8 Pediatric

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The HeaLMe post-market clinical follow-up registry is undertaken to evaluate the safety and performance of the index devices Heart Lung Machine HL 40 and Temperature Probes TPO-D-HLM L1.8 Adult / Pediatric in patients undergoing cardiac / thoracic / vascular surgery.

DETAILED DESCRIPTION:
In this study, patients who are connected to the index devices Heart Lung Machine HL 40 and Temperature Probes TPO-D-HLM L1.8 Adult / Pediatric and undergo a cardiac / thoracic / vascular surgery will be observed. This includes neonates, infants, adolescents and adults regardless of age and underlying health condition. It also includes elective, urgent and emergent surgeries.

Data will be collected for each participant according to the study schedule and standard routine clinical practice at the enrolling centers. There will be no additional visits, nor procedures pertaining to the study itself for subjects who participate in the study.

Informed consent of the patients will be obtained to allow the use of their clinical records for the purpose of this observational study before data are being collected.

The period of data collection for each patient will be only the index procedure. The index procedure is defined as the investigator's planned initial procedure in which the patient is connected to the HL 40 and the Temperature Probes. The index procedure starts with the cannulation of the patient for the index procedure and ends with the de-cannulation of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Signed Patient Informed Consent (including emergency approach)
* All patients who are connected to extracorporeal circulation using the index devices.

Exclusion Criteria:

* Pregnancy
* Current participation or planned participation in a concurrent drug or interventional medical device study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All eligible patients who are connected to the index devices and undergo a cardiac / thoracic / vascular surgery. This includes neonates, infants, adolescents and adults regardless of age and underlying health condition. It also includes elective, urgent and emergent surgeries.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Performance Endpoint | Only during the index procedure, no FU.
  The rate of cases performed by the index devices during the index procedure without any failure and / or malfunction related to the index device(s).
Safety Endpoint | Only during the index procedure, no FU.
  The rate of index device(s) related Adverse Events during the index procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Crespo de Hubsch, Dr., Principal Investigator — Hospital Universitario de Cruces
Locations (3):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy
- Spain (2):
  - Organización Sanitaria Integrada Ezkerraldea-Enkarterri-Cruces (Centro sanitario Hospital Universitario Cruces), Bilbao
  - Hospital Universitario Ramón y Cajal, Madrid

IPD SHARING:
Plan to Share IPD: No